CLINICAL TRIAL: NCT03092037
Title: Pharmacogenomics of Contraception: Genetic Variants and Etonogestrel Pharmacokinetics
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Other Study IDs: 16-2462
Record Dates: First submitted 2017-03-10; First posted 2017-03-27 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Contraception
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood samples will be collected at the enrollment visit and will undergo DNA extraction using commercial Qiagen® kits in Dr. Christina Aquilante's laboratory.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- All participants: All participants will have their blood drawn. DNA will be extracted from whole blood, and serum will be analyzed for ENG concentrations. Genotyping data will be analyzed for associations with serum ENG concentrations.
  Interventions: Procedure: Blood draw
- All participants (side-effects): All participants will have their blood drawn and complete a brief questionnaire regarding bleeding patterns and side-effects. DNA will be extracted from whole blood and genotyping data will be analyzed for associations with specific bleeding patterns and side-effects.
  Interventions: Procedure: Blood draw

INTERVENTIONS:
Procedure: Blood draw — The Investigators will collect serum and whole blood from participants.

SUMMARY:
The proposed study will investigate the relationship between genetic variants and serum contraceptive hormone levels, specifically the progestin etonogestrel. This study will provide the foundation for future pharmacogenomic investigations of more commonly used contraceptive methods with higher failure rates.

DETAILED DESCRIPTION:
Approximately 700 reproductive age women (18-45) with an Etonogestrel (ENG) contraceptive implant in place for more than 1 year will be enrolled. Participants will undergo a blood draw for measurement of ENG concentration (serum) and genotyping (whole blood) and complete a questionnaire regarding their demographics and contraceptive, gynecological, and obstetrical history. The research investigators will also consent participants for use of their genetic samples and clinical data in future unspecified research.

The serum samples will be de-identified for ENG analysis, which will be done using a liquid chromatography-mass spectrometry method. Additional whole blood samples collected at the enrollment visit will undergo DNA extraction. A candidate gene study was conducted using the first 350 participants. The research investigators selected 120 genetic variants for 14 target genes involved in progestin metabolism, regulation, and function for this candidate gene study. A Genome Wide Association Study will be performed using all 700 participants. Genotyping will be performed using a custom MultiEthnic Global Array chip through the Colorado Center for Personalized Medicine.

ELIGIBILITY:
Inclusion Criteria:

* women of reproductive age (18-45 years)
* have had an ENG contraceptive implant in place for 12-36 months

Exclusion Criteria:

* Use of medications or supplements in the past four weeks which could impact serum ENG levels through inhibition or induction of CYP enzymes (specifically CYP-3A4)
* Medical conditions that could impact baseline liver function (e.g. hepatitis, cirrhosis)
* Body mass index (BMI) less than 18.5

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Eligible participants must be females as we are studying the ENG contraceptive implant.
Study Population: We will enroll 900 women of reproductive age (18-45 years) who have had an ENG contraceptive implant in place for 12-36 months.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Actual)
Dates: Start 2017-03-23 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-04-29 (Actual)

PRIMARY OUTCOMES:
Proportion of genetic variants in cases versus controls | DNA extracted from whole blood specimens will be genotyped at the conclusion of enrollment, approximately 12 months.
  Genetic variants will be analyzed using a Taqman microarray chip for 120 pre-selected variants
Genome wide genotyping results | DNA extracted from whole blood specimens will be genotyped at the conclusion of enrollment, approximately 15 months.
  Participants will undergo genotyping using a custom MEGA chip at the Colorado Center for Personalized Medicine. Imputation of the chip results will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Lazorwitz, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lazorwitz A, Aquilante CL, Shortt JA, Gignoux CR, Teal S, Sheeder J. Pharmacogenomics of the Etonogestrel Contraceptive Implant: A Genome-Wide Association Study of Steady-State Etonogestrel Concentrations. O G Open. 2025 Feb 27;2(1):e066. doi: 10.1097/og9.0000000000000066. eCollection 2025 Feb. PMID 41000562
- [Derived] Lazorwitz A, Sheeder J, Teal S. The influence of lifestyle factors on serum etonogestrel concentrations among contraceptive implant users. Contraception. 2024 Dec;140:110539. doi: 10.1016/j.contraception.2024.110539. Epub 2024 Jul 11. PMID 39002624
- [Derived] Lazorwitz A, Sheeder J, Teal S. Variability in repeat serum etonogestrel concentrations among contraceptive implant users during the steady-release pharmacokinetic period. Contraception. 2022 Apr;108:65-68. doi: 10.1016/j.contraception.2021.12.008. Epub 2021 Dec 29. PMID 34973207
- [Derived] Lazorwitz A, Aquilante CL, Shortt JA, Sheeder J, Teal S, Gignoux CR. Applicability of ancestral genotyping in pharmacogenomic research with hormonal contraception. Clin Transl Sci. 2021 Sep;14(5):1713-1718. doi: 10.1111/cts.13014. Epub 2021 May 2. PMID 33650294
- [Derived] Lazorwitz A, Sheeder J, Teal S. An exploratory study on the association of lifestyle factors with serum etonogestrel concentrations among contraceptive implant users. Eur J Contracept Reprod Health Care. 2021 Aug;26(4):323-325. doi: 10.1080/13625187.2021.1887475. Epub 2021 Feb 17. PMID 33596152
- [Derived] Lazorwitz A, Aquilante CL, Sheeder J, Guiahi M, Teal S. Relationship between patient characteristics and serum etonogestrel concentrations in contraceptive implant users. Contraception. 2019 Jul;100(1):37-41. doi: 10.1016/j.contraception.2019.03.045. Epub 2019 Apr 10. PMID 30980827
- [Derived] Lazorwitz A, Aquilante CL, Oreschak K, Sheeder J, Guiahi M, Teal S. Influence of Genetic Variants on Steady-State Etonogestrel Concentrations Among Contraceptive Implant Users. Obstet Gynecol. 2019 Apr;133(4):783-794. doi: 10.1097/AOG.0000000000003189. PMID 30870275